CLINICAL TRIAL: NCT06574217
Title: Evaluation of Stepping Stones
Acronym: StSt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Policy & Research Group (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other); Public Health - Seattle and King County (Other Government); Reproductive Health National Training Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1 TP2AH000093-01-00
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Teen Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepping Stones (Experimental)
  Interventions: Behavioral: Stepping Stones (StSt)
- Like (Sham Comparator)
  Interventions: Behavioral: Like

INTERVENTIONS:
Behavioral: Stepping Stones (StSt) — StSt is an individual-level intervention designed to help youth make healthy decisions. StSt is delivered in-person by an adult guide during four ~30-50 minute sessions over a period of up to 8 weeks. The adult guide leads the youth through health-focused discussions related to identifying personal values, making a social network map, and then creating and refining individualized plans.
  Arms: Stepping Stones
Behavioral: Like — Like is an hour-long film that discusses the impact of social media on the brain. Study staff will organize for each individual participant to watch the film in-person. The film does not include information related to the outcomes of interest for the study.
  Arms: Like

SUMMARY:
The goal of this randomized trial is to learn if the Stepping Stones (StSt) intervention has a positive impact on the sexual health and relationship behaviors of sexually active youth between the ages of 12 and 22 years old who are at risk for or involved in the legal or child welfare systems. The primary research questions it aims to answer are:

* Three months after being offered the intervention, does StSt impact youth's receipt of sexually transmitted infection testing in the past four months?
* Nine months after being offered the intervention, does StSt impact youth's frequency of having vaginal and anal sex without condoms in the past four months?
* Nine months after being offered the intervention, does StSt impact youth's perpetration of emotional abuse in the past four months?

Researchers will compare participants randomized to receive StSt (treatment group) to participants randomized to receive a control condition that contains no sexual or reproductive health information (control group).

Participants randomized to the treatment group will be offered StSt as an-person, individual-based intervention delivered over four sessions during a 6-8 week period. Participants randomized to the control group will be offered a virtually delivered control condition.

DETAILED DESCRIPTION:
This is an individual-level, randomized control trial to rigorously evaluate the impact of the Stepping Stones (StSt) intervention. Participant outcomes will be assessed using self-reported, individual-level data gathered using a structured questionnaire administered at three time points: baseline (enrollment); three months post-intervention (five months after baseline); and nine months post-intervention (eleven months after baseline).

ELIGIBILITY:
Inclusion Criteria:

* At risk for or involved in the legal or child welfare systems
* Report ever having vaginal and/or anal sex and plan to have sex in the next six months
* Comfortable reading, speaking, and writing in English

Exclusion Criteria:

* Currently trying to start a pregnancy
* Currently in jail or being detained in a facility
* Enrolled in an ongoing PRG-run TPP study
* Identified as fraudulent (only for individuals recruited online)

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Identifies as male or non-binary gender
Enrollment: 650 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-09-14 (Estimated)

PRIMARY OUTCOMES:
Receipt of sexually transmitted infection (STI) testing in the past four months | Assessed three months after the intervention period has ended (five months post-baseline)
  Participants are asked the following item:
  1) Have you been tested for sexually transmitted infections (STIs) in the past 4 months? The resulting variable is dichotomous with values 0 or 1, where 0 indicates a person who has not received STI testing in the past four months and 1 indicates a person who has received STI testing in the past four months.
Times having vaginal and anal sex without condoms in the past four months | Assessed nine months after the intervention period has ended (eleven months post-baseline)
  Participants are asked the following two items:
  1. In the past 4 months, how many times have you had vaginal sex without you or your sexual partner using a condom?
  2. In the past 4 months, how many times have you had anal sex without you or your sexual partner using a condom? The resulting variable is continuous with values that range from 0 to k, where 0 indicates that a person has not engaged in vaginal and anal sex without a condom in the past four months, and k indicates the number of times the person has engaged in vaginal and anal sex without a condom in the past four months.
Perpetration of emotional abuse | Assessed nine months after the intervention period has ended (eleven months post-baseline)
  Participants are asked how many times in the past four months they have done the following things to a sexual or romantic partner:
  1. Damaged something on purpose that belonged to them?
  2. Said things to hurt their feelings on purpose?
  3. Insulted them in front of others?
  4. Would not let them talk to or do things with other people?
  5. Threatened to start dating someone else?
  6. Did something just to make them jealous?
  7. Blamed them for bad things you did?
  8. Threatened to hurt them?
  9. Made them report where they were every minute of the day?
  10. Put down their looks?
  11. Threw something at them but missed?
  12. Told them they could not talk to someone else?
  13. Started to hit them but stopped?
  14. Brought up something from the past to hurt them? Participants are provided with four response options: 0 times; 1 to 3 times; 4 to 9 times; or 10 or more times.
  The measure is calculated as the average response to all 14 items in the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Walsh, Ph.D., Principal Investigator — The Policy & Research Group
Locations (1):
- The Policy & Research Group, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A dataset will be prepared at the conclusion of the study, which includes deidentified individual-level data on all study participants who contributed self report data. Respondents will be represented only by a research ID number. Included in the dataset will be self-report data collected across all survey administrations (including demographic characteristics, sexual behaviors, and theoretical antecedents to those behaviors) and select information on program participation (e.g., which program components were completed). Basic data cleaning steps will be taken in order to ensure data are unidentifiable and to increase usability.
Supporting Information: SAP
Time Frame: The individual participant dataset will become available twelve months after the study has concluded.